CLINICAL TRIAL: NCT00217789
Title: Pathogen Specific Immunity in Sarcoidosis
Brief Title: Pathogen Specific Immunity in Patients With Sarcoidosis
Status: Completed | Type: Observational
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Other Study IDs: 0120040230; M-230-2004; 287; R21HL077462-02 (NIH); R21HL077462 (NIH)
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis | interventions — Bronchoalveolar Lavage; Phlebotomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Bronchoalveolar Lavage and Venipuncture

SUMMARY:
The purpose of this study is to assess the lung cells of healthy volunteers and patients with stage II and III pulmonary sarcoidosis for pathogen specific memory immunity and gene expression patterns.

DETAILED DESCRIPTION:
BACKGROUND:

Since its initial description 125 years ago, sarcoidosis continues to be a "challenging" disease. Its etiology remains unknown. Discovering the etiology of sarcoidosis remains a major goal with important implications regarding treatment, predicting outcome, as well as determining approaches for preventive measures. Immunological responses and granulomatous tissue formation characterizing sarcoidosis are similar to those observed in a variety of infectious diseases. However, the nature of the specific antigen(s), which putatively trigger the inflammatory response in sarcoidosis, remains elusive. Occurrence of sarcoidosis in spatially related clusters, and household and health care settings strongly support person-to-person transmission of an infectious agent as one of the potential causes of this disease. Sarcoidosis has been associated with a variety of infectious agents, none of which can be cultured. Propionibacterium acnes (P. acnes) and M.tuberculosis (Mtb) are the most commonly identifiable infectious pathogens by PCR-based methods and considered to be associated with the development of this disease. Immunological studies in sarcoidosis have focused largely on the assessment of constitutive, immune responses and the description of the phenotypes of blood and lung cells in patients and control subjects.

DESIGN NARRATIVE:

This study will utilize memory immune responses as search tools for the 'immunological imprints' from P. acnes or Mtb exposure. Peripheral blood mononuclear cells and bronchoalveolar cells will be compared from patients with stage II and/or stage III sarcoidosis and from healthy control subjects. Investigators will use ELISPOT assay to study: (1) frequencies of pathogen-specific interferon-7 and interleukin-10-producing cells, and (2) utilizing P. acnes- or Mtb-infected autologous monocytes and alveolar macrophages as target cell frequencies of pathogen-specific granzyme B-releasing cytotoxic T lymphocytes and natural killer cells. Finally, investigators will test the feasibility of identifying by DNA micro array, pathogen specific, transcriptional host gene expression profiles in P. acnes- and Mtb-stimulated blood cells from healthy control subjects and patients with active sarcoidosis and to compare these with gene expression profiles from autologous, unstimulated in situ lung cells. The studies will address the role of P. acnes and Mtb in the etiology of sarcoidosis and will also serve as a basis or model for future work involving other possible infectious or non-infectious pathogens/antigens for the development of sarcoidosis.

ELIGIBILITY:
Inclusion Criteria for Sarcoidosis Participants:

* Clinical and radiographic signs and symptoms consistent with pulmonary sarcoidosis stage II or III and confirmed histopathology
* No prior corticosteroid or immune suppressive or immune modulating therapies

Inclusion Criteria for Healthy Participants:

* No clinical and radiographic signs and symptoms of respiratory or other chronic or systemic illness

Exclusion Criteria for All Participants:

* Unwilling or unable to provide informed consent
* Unwilling or unable to comply with all study requirements
* History of upper or lower respiratory tract infection within 1 month of study entry
* History of major occupational or microbial exposures known to be associated with granulomatous inflammatory responses
* Positive HIV-1 serology
* Severe psychiatric disease
* Cough-induced syncope
* History of massive hemoptysis or history of pneumothorax, tuberculosis, and immunosuppressive therapies
* Presence of any chronic medical condition requiring daily medication
* Gingivitis or other infectious processes in the oral cavity
* Positive skin test to purified protein derivative (tuberculin)
* Hemoglobin level less than 10g/dl
* Illicit drug use or history of cigarette smoking within 1 year prior to study entry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sarcoidosis patients and healthy subjects
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2004-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Pathogen Specific Immunity in Sarcoidosis | July 2004 - June 2008
  Toxicity, DEP-Induced Cytokines, Effect of DEP on Stimulant-Induced Cytokine Production, in vitro Effects of DEP on M.tb-induced Cytokine Production, time kinetics of In vitro effects of DEP on M.tb-induced cytokine production, effect of DEP Exposure on M.tb H37Ra-induced Lymphocyte Proliferation, whole blood killing experiments

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Schwander, MD, PhD, Principal Investigator — University of Medicine and Dentistry of New Jersey
Locations (1):
- University of Medicine and Dentistry of New Jersey, Newark, New Jersey, United States